CLINICAL TRIAL: NCT05915546
Title: A Phase 1, Open-label Trial to Evaluate the Effect of Food on the Pharmacokinetics of Emraclidine in Healthy Adult Participants
Brief Title: The Effect of Food on the Pharmacokinetics (PK) of Emraclidine in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CVL-231-HV-1009
Record Dates: First submitted 2023-06-13; First posted 2023-06-23 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Emraclidine (Fasted then Fed) (Experimental): Single oral dose of Emraclidine 15 mg tablet under fasted (without food) condition followed by fed condition in treatment period 1 and 2, respectively.
  Interventions: Drug: Emraclidine
- Emraclidine (Fed then Fasted) (Experimental): Single oral dose of Emraclidine 15 mg tablet under fed condition followed by fasted (without food) condition in treatment period 1 and 2, respectively.
  Interventions: Drug: Emraclidine

INTERVENTIONS:
Drug: Emraclidine — Tablets

SUMMARY:
The primary purpose of this study is to evaluate the effect of food (a high-fat meal) on the pharmacokinetics of emraclidine and metabolite CV-0000364 following single oral dose administration in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female (both women of childbearing and nonchildbearing potential) participants, ages 18 to 55 years, at the time of signing the informed consent form (ICF).
2. Sexually active women of childbearing potential must agree to use an acceptable birth control method, during the trial and for 7 days after the last dose. Acceptable birth control methods that result in a failure rate of more than 1% per year include the following:

   * Progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action
   * Male or female condom with or without spermicide
   * Cap, diaphragm, or sponge with spermicide
3. Body mass index of 17.5 to 32.0 kilograms per square meter (kg/m^2), inclusive, and total body weight >45 kg (110 pounds [lb]) at Screening.
4. Healthy as determined by medical evaluation, including medical and psychiatric history, physical and neurological examinations, ECG, vital sign measurements, and laboratory test results, as evaluated by the investigator.
5. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the full protocol.
6. Ability, in the opinion of the investigator, to understand the nature of the trial and comply with protocol requirements, including the prescribed dosage regimens, scheduled visits, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Current or past history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, genitourinary, endocrine (including diabetes mellitus, thyroid disorders), malignancy, hematological, immunological, neurological, or psychiatric disease that, in the opinion of the investigator or medical monitor, could compromise either participant safety or the results of the trial.
2. "Yes" responses for any of the following items on the C-SSRS (within the individual's lifetime):

   * Suicidal Ideation Item 3 (Active Suicidal Ideation With Any Methods [Not Plan] Without Intent to Act)
   * Suicidal Ideation Item 4 (Active Suicidal Ideation With Some Intent to Act, Without Specific Plan)
   * Suicidal Ideation Item 5 (Active Suicidal Ideation With Specific Plan and Intent)
   * Any of the Suicidal Behavior items (Actual Attempt, Interrupted Attempt, Aborted Attempt, or Preparatory Acts/Behavior) "Yes" responses for any of the following items on the C-SSRS (within past 12 months):
   * Suicidal Ideation Item 1 (Wish to be Dead)
   * Suicidal Ideation Item 2 (Non-Specific Active Suicidal Thoughts) Serious risk of suicide in the opinion of the investigator is also exclusionary
3. Any condition or surgery that could possibly affect drug absorption, including, but not limited to, bowel resections, bariatric weight loss surgery/procedures, gastrectomy, and cholecystectomy.
4. Use of any prescription and over-the-counter medications from 28 days prior to first dose of Investigational Medical Product or likely to require concomitant therapy (e.g., prescription and over-the counter medications, herbal medications, vitamins, and supplements) during the trial, with the exception of acetaminophen (maximum total daily dose of 2 g) and topical hydrocortisone as needed for treatment of an Adverse Event(AE). Vaccinations or boosters within 7 days of planned dosing or while on trial are prohibited.
5. Positive result for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody with detectable viral ribonucleic acid (RNA) levels at Screening.
6. Positive drug screen or a positive test for alcohol at Screening or Baseline Visits.
7. Female participants who are pregnant, breastfeeding, or planning to become pregnant during IMP treatment or within 7 days after the last dose of IMP. Women of childbearing potential must have a negative serum pregnancy test result at the Screening Visit and a negative urine pregnancy test result at baseline.
8. Any of the following clinical laboratory test results at the Screening Visit (as assessed by the central laboratory) and at Check-in (Day -1; as assessed by the local laboratory), and confirmed by a single repeat measurement, if deemed necessary:

   * aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2.0 × upper limit normal (ULN)
   * Total bilirubin >1.5 × ULN. If Gilbert's syndrome is suspected, total bilirubin >1.5 × ULN is acceptable if the conjugated or direct bilirubin fraction is <20% of total bilirubin.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Emraclidine and its Metabolite CV-0000364 | Pre-dose and at multiple timepoints up to Day 6
Time to Maximum Plasma Concentration (Tmax) of Emraclidine and its Metabolite CV-0000364 | Pre-dose and at multiple timepoints up to Day 6
Area Under the Plasma Concentration-time Curve from Time Zero to Last Specified Sampling Time (AUC0-t) of Emraclidine and its Metabolite CV-0000364 | Pre-dose and at multiple timepoints up to Day 6
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUCinf) of Emraclidine and its Metabolite CV-0000364 | Pre-dose and at multiple timepoints up to Day 6

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to Day 13
Number of Participants With Clinically Significant Changes in Vital Sign Measurements | Up to Day 13
Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Parameters | Up to Day 13
Number of Participants With Clinically Significant Changes in Laboratory Assessments | Up to Day 13
Number of Participants With Clinically Significant Changes in Physical and Neurological Examination Results | Up to Day 13
Changes in Suicidality Assessed Using the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to Day 13
  The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe). Greater lethality or potential lethality of suicidal behaviors (endorsed on the behavior subscale) indicates increased risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Dilworth, Minnesota, Dilworth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No